CLINICAL TRIAL: NCT06447025
Title: Jive: An Open Label Extension Study to Assess the Long-term Safety, Efficacy, Pharmacodynamics, Pharmacokinetics, and Tolerability of Subcutaneous CTI-1601 in Subjects With Friedreich's Ataxia
Brief Title: An Open Label Extension Study of CTI-1601 in Subjects With Friedreich's Ataxia
Acronym: Jive
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Larimar Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-1601-201
Record Dates: First submitted 2024-02-15; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTI-1601 (Experimental): CTI-1601 will be administered daily
  Interventions: Biological: CTI-1601

INTERVENTIONS:
Biological: CTI-1601 — CTI-1601 is a recombinant fusion protein and is intended to deliver human frataxin, the protein deficient in Friedreich's ataxia
  Other Names: Nomlabofusp

SUMMARY:
This is an open-label extension (OLE) study designed to evaluate the long-term safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and clinical effects of subcutaneous (SC) administration of CTI-1601, also known as nomlabofusp, in subjects with Friedreich's ataxia (FRDA).

The objectives of this OLE study are:

* To evaluate the safety of long-term subcutaneous (SC) administration of CTI-1601 in subjects with FRDA
* To evaluate the PK of long-term subcutaneous (SC) administration of CTI-1601 in subjects with FRDA
* To evaluate the effect of long-term subcutaneous (SC) administration of CTI-1601 in subjects with FRDA on:

  * Tissue FXN concentrations
  * Clinical evaluations of FRDA
  * Gene Expression and select lipids

DETAILED DESCRIPTION:
This is an open label extension (OLE) study in patients with FRDA who participated in a prior clinical study of CTI-1601 to evaluate the safety, PK, PD, and clinical effects of long-term daily administration of CTI-1601.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with FRDA who previously completed participation in a study of CTI-1601 will be eligible to participate in this study unless the subject experienced one or more of the following in a previous CTI-1601 study: a) serious adverse event (SAE) related to study drug; b) significant AE, defined as Grade 3 or higher according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 (or higher), related to study drug; c) some other event, related to participation in a previous study with CTI-1601, that supports the exclusion of the subject from participating in this study as determined by the Sponsor (i.e., an AE considered clinically significant by the Sponsor regardless of whether it met SAE criteria and regardless of CTCAE grade); d) Withdraw from participation in a previous study of CTI-1601 for any reason.
* Subject has a HbA1c less than or equal to 7.0%.
* Subject must demonstrate sufficient dexterity and visual acuity to prepare and self-administer SC injections of CTI-1601 QD or is able to identify a caregiver who will be trained and committed to prepare and administer the daily injections.

Exclusion Criteria:

Subjects are excluded from the study if any of the following exclusion criteria are met:

* Subjects who are confirmed as compound heterozygous (GAA repeat expansion on only one allele) for FRDA.
* Subject has any condition, disease, or situation, including a cardiac condition or disease, that in the opinion of the PI, could confound the results of the study or put the subject at undue risk, making participation inadvisable.
* Subject used any investigational drug (other than CTI-1601) or device within 90 days prior to Screening.
* Subject requires use of amiodarone.
* Subject used erythropoietin, etravirine, or gamma interferon within 90 days prior to Screening.
* Subject use of biotin supplementation that exceeds 30 mcg/day, either as part of a multivitamin or as a standalone supplement, within 7 days prior to the first dose of study drug. Biotin supplementation ≤30 mcg/day is permitted if taken at a stable dose and frequency for at least 28 days prior to Screening and there is a commitment from the subject to maintain the biotin dose throughout the study (due to interference with assays).
* Subject uses more than 3 grams of acetaminophen daily.
* Subject receives medication that requires SC injection in the abdomen or thigh.
* Subject is unable to discontinue medications that have not been at a stable dose and frequency for at least 28 days prior to Screening.
* Subject has a Screening echocardiogram (ECHO) LVEF < 45%.
* Male subject has a QTcF > 450 milliseconds or female subject has a QTcF > 470 milliseconds on an ECG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with treatment-emergent adverse events (TEAEs) by System Organ Class (SOC), Preferred Term (PT) and Maximum Severity | Up to 24 months
Number of subjects with abnormal laboratory test results | Up to 24 months
Change from baseline in electrocardiogram (ECG) parameters including, but not limited to, HR, RR interval, PR interval, QRS duration, QT interval, and QTcF interval | Up to 24 months
Change from baseline in left ventricular ejection fraction (LVEF) | Up to 24 months
  LVEF indicates the percentage of change in LV volume from diastole to systole that measures how well the left ventricle of the heart pumps blood.
Change from baseline in left ventricular end-diastolic volume (LVEDV) | Up to 24 months
  LVEDV is the amount of blood, measured in milliliters (mL), in the heart's left ventricle just before the heart contracts.
Change from baseline in blood pressure (mmHg) | Up to 24 months
Change from baseline in pulse (bpm) | Up to 24 months
Change from baseline in temperature (°C) | Up to 24 months
Change from baseline in respiration rate (breaths per minute) | Up to 24 months
Number of subjects with any suicidal ideation or behavior (Categories 1-10) of the Columbia Suicide Severity Rating Scale (C-SSRS) | Up to 24 months
  The Columbia Suicide Severity Rating Scale (C-SSRS) is a tool used to assess the occurrence, severity, and frequency of suicidal thoughts and behaviors. A higher score on the C-SSRS generally indicate a worse outcome, as they signify a higher level of suicidal ideation or behavior.
Change from baseline at each collection timepoint in tissue frataxin concentrations normalized to total protein observed in buccal cells collected from cheek swabs and skin cells collected from skin punch biopsies | Up to 24 months
Change from baseline in motor function as assessed by 9-hole peg test (9-HPT) | Up to 24 months
Change from baseline in motor function as assessed by the timed 25-foot walk test (T25-FW) | Up to 24 months
Change from baseline in neurologic function as assessed by the modified Friedreich's Ataxia Rating Scale (mFARS) total score | Up to 24 months
  The Modified Friedreich's Ataxia Rating Scale (mFARS) is a modified neurologic scale involving direct subject participation and targets specific areas impacted by Friedreich's ataxia (bulbar, upper limb, lower limb, and upright stability), with scores ranging from 0-67 points, with higher scores indicating a greater level of disability.
Change from baseline in neurologic function as assessed by the upright stability subscale examination of the mFARS | Through study completion, up to 24 months
  The Upright Stability Subscale is an assessment of an individual's ability to maintain balance and stability while standing upright. It has a minimum value of 0 and a maximum value of 36. A higher score indicates a better outcome, reflecting greater stability and balance abilities while standing upright.
Change in activities of daily living (ADLs) as assessed by the Friedreich's Ataxia Rating Scale Activities of Daily Living (FARS_ADL) | Up to 24 months
  The FARS_ADL, scored 0 to 36, is a subscale of FARS assessing a subject's ability to complete activities of daily living. A higher score indicates a greater level of disability. The FARS_ADL questionnaire will be performed at the timepoints indicated in protocol.
Change from baseline in total fatigue score and all the subscale scores as assessed by the Fatigue Impact Scale (MFIS) | Up to 24 months
  The Modified Fatigue Impact Scale (MFIS) is a revised form of the Fatigue Impact Scale based on items derived from interviews with MS patients concerning how fatigue impacts their lives. This instrument provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. Participants rate on a 5-point scale, with 0 = 'Never' to 4 = 'Almost always' their agreement with 21 statements. Total score (0-84) and subscales for physical (0-36), cognitive (0-40) and psychosocial functioning (0-8). The 5-item version is scored (0-20). Higher numbers indicate greater fatigue. The MFIS will be performed at the timepoints indicated in protocol.
Change from baseline in the assessment of disease as assessed by the Functional Staging for Ataxia | Up to 24 months
Overall impression of change as assessed by the patient using the Patient Global Impression of Change (PGI-C) Scale | Up to 24 months
  The Patient Global Impression of Change (PGI-C) reflects a patient's assessment about the efficacy of treatment. PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse." The PGI-C will be performed at the timepoints indicated in protocol.
Overall impression of change assessed by a clinician using the Clinical Global Impression of Change (CGI-C) | Up to 24 months
  The Clinical Global Impression of Change (CGI-C) is an assessment to measure change in clinical status (symptoms and functional ability) of the subject's condition from baseline with study drug. CGI-C scores range from 1 (very much improved) through to 7 (very much worse). The CGI-C will be performed at the timepoints indicated in protocol.
Area under the concentration-time curve for the dosing interval (AUC0-tau) | Days 1, 30, 60, 90: pre-dose, 5, 15, 30 minutes after the dose, and 1, 2, 4, 6, 8 hours after the dose; Day 180: pre-dose and 5, 15 minutes after the dose; Days 270, 360, Q3M thereafter: pre-dose; through study completion, up to 24 months
Area under the concentration-time curve from time 0 to the time of last quantifiable concentration (AUC0-t) | Days 1, 30, 60, 90: pre-dose, 5, 15, 30 minutes after the dose, and 1, 2, 4, 6, 8 hours after the dose; Day 180: pre-dose and 5, 15 minutes after the dose; Days 270, 360, Q3M thereafter: pre-dose; through study completion, up to 24 months
Mean maximum observed concentration (Cmax) | Days 1, 30, 60, 90: pre-dose, 5, 15, 30 minutes after the dose, and 1, 2, 4, 6, 8 hours after the dose; Day 180: pre-dose and 5, 15 minutes after the dose; Days 270, 360, Q3M thereafter: pre-dose; through study completion, up to 24 months
Mean time of maximum observed concentration (Tmax) | Days 1, 30, 60, 90: pre-dose, 5, 15, 30 minutes after the dose, and 1, 2, 4, 6, 8 hours after the dose; Day 180: pre-dose and 5, 15 minutes after the dose; Days 270, 360, Q3M thereafter: pre-dose; through study completion, up to 24 months
Concentration reached immediately before the next dose is administered (Ctrough) | Days 1, 30, 60, 90: pre-dose, 5, 15, 30 minutes after the dose, and 1, 2, 4, 6, 8 hours after the dose; Day 180: pre-dose and 5, 15 minutes after the dose; Days 270, 360, Q3M thereafter: pre-dose; through study completion, up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Larimar Therapeutics, Inc., Study Chair — Larimar Therapeutics, Inc.
Locations (7):
- United States (7):
  - University of California Los Angeles, Los Angeles, California
  - Fixel Institute for Neurological Disease, University of Florida Health, Gainesville, Florida
  - Morsani Center for Advanced Health Care, University of South Florida Health, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - Clinilabs Drug Development, Corp., Eatontown, New Jersey
  - Ohio State University United States, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delatycki MB, Corben LA. Clinical features of Friedreich ataxia. J Child Neurol. 2012 Sep;27(9):1133-7. doi: 10.1177/0883073812448230. Epub 2012 Jun 29. PMID 22752493
- [Background] Deutsch EC, Santani AB, Perlman SL, Farmer JM, Stolle CA, Marusich MF, Lynch DR. A rapid, noninvasive immunoassay for frataxin: utility in assessment of Friedreich ataxia. Mol Genet Metab. 2010 Oct-Nov;101(2-3):238-45. doi: 10.1016/j.ymgme.2010.07.001. Epub 2010 Jul 8. PMID 20675166
- [Background] Fahey MC, Corben L, Collins V, Churchyard AJ, Delatycki MB. How is disease progress in Friedreich's ataxia best measured? A study of four rating scales. J Neurol Neurosurg Psychiatry. 2007 Apr;78(4):411-3. doi: 10.1136/jnnp.2006.096008. Epub 2006 Oct 20. PMID 17056635
- [Background] Fisk JD, Ritvo PG, Ross L, Haase DA, Marrie TJ, Schlech WF. Measuring the functional impact of fatigue: initial validation of the fatigue impact scale. Clin Infect Dis. 1994 Jan;18 Suppl 1:S79-83. doi: 10.1093/clinids/18.supplement_1.s79. PMID 8148458
- [Background] Goodkin DE, Hertsgaard D, Seminary J. Upper extremity function in multiple sclerosis: improving assessment sensitivity with box-and-block and nine-hole peg tests. Arch Phys Med Rehabil. 1988 Oct;69(10):850-4. PMID 3178453
- [Background] Koeppen AH. Friedreich's ataxia: pathology, pathogenesis, and molecular genetics. J Neurol Sci. 2011 Apr 15;303(1-2):1-12. doi: 10.1016/j.jns.2011.01.010. PMID 21315377
- [Background] Guidelines MSCfCP. Fatigue and multiple sclerosis: evidence-based management strategies for fatigue in multiple sclerosis. 1998.
- [Background] Lazaropoulos M, Dong Y, Clark E, Greeley NR, Seyer LA, Brigatti KW, Christie C, Perlman SL, Wilmot GR, Gomez CM, Mathews KD, Yoon G, Zesiewicz T, Hoyle C, Subramony SH, Brocht AF, Farmer JM, Wilson RB, Deutsch EC, Lynch DR. Frataxin levels in peripheral tissue in Friedreich ataxia. Ann Clin Transl Neurol. 2015 Aug;2(8):831-42. doi: 10.1002/acn3.225. Epub 2015 Jul 1. PMID 26339677
- [Background] Pandolfo M. Friedreich ataxia. Arch Neurol. 2008 Oct;65(10):1296-303. doi: 10.1001/archneur.65.10.1296. PMID 18852343
- [Background] Rudick R, Antel J, Confavreux C, Cutter G, Ellison G, Fischer J, Lublin F, Miller A, Petkau J, Rao S, Reingold S, Syndulko K, Thompson A, Wallenberg J, Weinshenker B, Willoughby E. Clinical outcomes assessment in multiple sclerosis. Ann Neurol. 1996 Sep;40(3):469-79. doi: 10.1002/ana.410400321. PMID 8797541
- [Background] Wang C, Lu N, Chen WC, Li H, Tiwari R, Xu Y, Yue LQ. Propensity score-integrated composite likelihood approach for incorporating real-world evidence in single-arm clinical studies. J Biopharm Stat. 2020 May 3;30(3):495-507. doi: 10.1080/10543406.2019.1684309. Epub 2019 Nov 10. PMID 31707908